CLINICAL TRIAL: NCT04518553
Title: Shanghai Pudong Hospital
Brief Title: Plasma Purification and Chronic Hepatitis B
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Pudong Hospital (Other)
Responsible Party: Principal Investigator, Jin HM, MD, professor, Shanghai Pudong Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ShanghaiPudongH4
Record Dates: First submitted 2020-08-11; First posted 2020-08-19 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2020-08

CONDITIONS: Chronic Hepatitis b
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active control (Active Comparator): antiviraltherapy using HA using antiviralHA drugs of HA to decrease HBV-DNA load. In this group, patients with chronic hepatitis B just take antiviral drug of HAs to control hepatitis B viral without active interference.
  Interventions: Drug: active comarator using antiviral drug of nucleoside analogues
- active interference (Experimental): HA+plasma purification as active interference. HA antiviral therapy using HA plus plasma purification every three months.DFT as plasma purification mode will be used. DFT therapy time lasts 2.5-3 hours each time.After three months, DFT therapy will be used if patients' HBV-DNA loads are higher than cut-off normal level.
  Interventions: Device: HA+purification

INTERVENTIONS:
Drug: active comarator using antiviral drug of nucleoside analogues — using antiviral drug of nucleoside analogues without additional active interference to control Hepatitis B virus.
  Arms: active control
Device: HA+purification — Based on antiviral drug of nucleoside analogues, plasma purification is added to control hepatitis B virus every three months. After three months, plasma purification will continue if hepatitis B virus DNA titer is still higher than cut-off normal value. plasma purification process lasts 2.5-3 hours each session.
  Arms: active interference

SUMMARY:
To compare the efficacy of nucleoside analogues （HA） alone and plasma purification +HA in reducing HBV viral load.

DETAILED DESCRIPTION:
Chronic hepatitis B (CHB) is a major disease harmful to human health and an important cause of liver cirrhosis and liver cancer. Hepatitis B virus (HBV) cccDNA exists for a long time in the liver of infected persons and serves as a template for HBV replication, which makes it difficult to eradicate HEPATITIS B virus infection. Antiviral drugs are commonly used clinically, including interferon and nucleoside analogues, but there are problems of recurrence and drug resistance. These drugs are not directly targeted at cccDNA and are therefore inefficient at reducing cccDNA. How to quickly and efficiently reduce the viral load of HBV-DNA, inhibit THE TRANSCRIPTION of HBV-CCCDNA RNA, and promote the negative conversion of HBeAg is an urgent problem to be solved at present, so it is particularly important to find other more effective drugs or methods. Plasma purification is a new treatment method in which the pathogenic factors (hepatitis B virus, etc.) are trapped in the hollow fibers by special membrane materials and removed. Therefore, this study adopts the randomized control method to explore the effect of plasma purification on HBV clearance, aiming to explore the effectiveness and safety of plasma purification in reducing HBV DNA viral load and inhibiting HBV cccDNA RNA transcription, so as to provide new treatment ideas and methods for future treatment of hepatitis B virus infection, which is beneficial to the society and individuals.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of Chronic hepatitis B Disease
2. hepatitis B virus HBeAg is positive
3. hepatitis B virus HBV-DNA virus load is more than 100000cps/ml

Exclusion Criteria:

1. Hypotension
2. Cardiopulmonary insufficiency
3. Coagulation disorders
4. Heparin allergy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2021-03-23 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Concentration of HBV(hepatitis B virus) HBeAg is serologically negative | 2 years
  serological examination every three months

SECONDARY OUTCOMES:
Concentration of HBV-DNA virus load is undetected | 2 years
  serological examination by compared of HAs with HAs+plasma purification treatment
Concentration of hepatitis B virus cccDNA RNA transcription becomes undetectedly | 2 years
  serological examination every three months
hepatitis B virus HBsAg serological transformation is negative | 2 years
  serological examination every three months

CONTACTS AND LOCATIONS:
Overall Officials: Hui Min Jin, MD, Principal Investigator — Fudan University

IPD SHARING:
Plan to Share IPD: No